CLINICAL TRIAL: NCT00949650
Title: A Randomised, Open-label, Phase III Study of BIBW 2992 Versus Chemotherapy as First-line Treatment for Patients With Stage IIIB or IV Adenocarcinoma of the Lung Harbouring an EGFR Activating Mutation
Brief Title: BIBW 2992 (Afatinib) Versus Chemotherapy as First Line Treatment in NSCLC With EGFR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.32; 2008-005615-18 (EudraCT Number)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — Pemetrexed; Afatinib; Cisplatin

ARMS (2):
- BIBW 2992 (Experimental): BIBW 2992 tablet once daily until progression
  Interventions: Drug: BIBW 2992
- Cisplatin/Pemetrexed (Active Comparator): Cisplatin and Pemetrexed IV once every 3 weeks for up to 6 cycles
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed IV given once every 3 weeks for up to 6 cycles
  Arms: Cisplatin/Pemetrexed
Drug: BIBW 2992 — BIBW 2992 once daily until progression
  Arms: BIBW 2992
Drug: Cisplatin — Cisplatin IV given once every 3 weeks for up to 6 cycles
  Arms: Cisplatin/Pemetrexed

SUMMARY:
This randomised, open label phase III trial will be performed in patients with adenocarcinoma of the lung with tumours harbouring an Epidermal Growth Factor Receptor activating mutation. The objectives of the trial are to compare the efficacy of single agent BIBW 2992, Arm A, with Pemetrexed/Cisplatin chemotherapy, Arm B, as first line treatment for this group of patients.

ELIGIBILITY:
Inclusion criteria:

* Pathologically confirmed diagnosis of Stage IIIB (with cytologically proven pleural effusion or pericardial effusion) or Stage IV adenocarcinoma of the lung. Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Epidermal Growth Factor Receptor mutation detected by central laboratory analysis of tumour biopsy material.
* Measurable disease according to RECIST 1.1.
* Eastern Cooperative Oncology Group score of 0 or 1.
* Age >/= 18 years.
* Life expectancy of at least three months.
* Written informed consent that is consistent with International Conference on Harmonisation-Good Clinical Practice guidelines.

Exclusion criteria:

* Prior chemotherapy for relapsed and/or metastatic NSCLC. Neoadjuvant/adjuvant chemotherapy is permitted if at least 12 months has elapsed between the end of chemotherapy and randomisation.
* Prior treatment with Epidermal Growth Factor Receptor targeting small molecules or antibodies.
* Radiotherapy or surgery (other than biopsy) within 4 weeks prior to randomisation.
* Active brain metastases
* Any other current malignancy or malignancy diagnosed within the past five years
* Known pre-existing interstitial lung disease.
* Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom.
* History or presence of clinically relevant cardiovascular abnormalities.
* Any other concomitant serious illness or organ system dysfunction.
* Adequate absolute neutrophil count and platelet count
* Adequate liver and kidney function
* Active hepatitis B infection, active hepatitis C infection or known HIV carrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2009-08-14 (Actual); Primary Completion 2012-02-09 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (133):
- United States (7):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Clinical Trials and Research Associates Inc, Montebello, California
  - Innovative Medical Research of South Florida, Miami, Florida
  - Crescent City Research Consortiom, Marrero, Louisiana
  - Interlakes Foundation, Incorporated, Rochester, New York
  - Lehigh Valley Hospital / Lehigh Valley Health Network, Allentown, Pennsylvania
  - South Texas Institute of Cancer, Northwest Cancer Center, Corpus Christi, Texas
- Argentina (8):
  - Instituto de Medicina Nuclear de Bahía Blanca, Bahía Blanca
  - Hospital Alemán, Capital Federal
  - Imcaba S.R.L., Capital Federal
  - IMAI Research, Capital Federal
  - Instituto Alexander Fleming, Capital Federal
  - Hospital Militar Central, Capital Federal
  - PALIAR, Capital Federal
  - Centro Oncológico de Rosario, Rosario
- Australia (9):
  - Lifehouse, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Burnside War Memorial Hospital, Toorak Gardens, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St. Vincents Hospital (MEL), Fitzroy, Victoria
  - Mount Medical Centre, Perth, Western Australia
- Austria (3):
  - KH d. Elisabethinen Linz, Linz
  - SMZ Baumgartner Hoehe Otto Wagner Spital, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (5):
  - Brussels - UNIV St-Pierre, Brussels
  - UNIV UZ Gent, Ghent
  - Brussels - UNIV UZ Brussel, Jette
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (5):
  - Centro de Pesquisa do Hospital Lifecenter, Belo Horizonte
  - Centro de Pesquisas Clínicas em Oncología, Cachoeiro de Itapemirim
  - Insituto de Oncologia do Paraná, Curitiba
  - Hospital São Lucas da Pontifícia Universidade Católica, Porto Alegre
  - UNIFESP Departamento de Medicina de Pneumologia, São Paulo
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute (University of Alberta), Edmonton, Alberta
  - Charles LeMoyne Hospital, Greenfield Park, Migration Data
  - Hematologiste et oncologue medical CHUM - Hopital Notre-Dame, Montreal, Migration Data
  - McGill University, Department of Oncology, Montreal, Migration Data
- Chile (3):
  - Hospital Dirección de Previsión de Carabineros, Los Condes
  - Instituto Oncológico Limitada Viña del Mar, Reñaca
  - Instituto Clínico Oncológico del Sur - ICOS, Temuco
- France (9):
  - HOP d'Angers, Angers
  - HOP Côte de Nacre, Caen
  - HOP Nord Michallon, La Tronche
  - HOP Croix Rousse, Pneumo, Lyon, Lyon
  - INS Curie, Paris
  - HOP Sud-Réunion, Pneumo, Saint Pierre, Saint Pierre - La Réunion
  - CTR René Gauducheau, Saint-Herblain
  - HOP - HIA Sainte Anne, Toulon
  - HOP, Pneumo, Villefranche sur Saône, Villefranche-sur-Saône
- Germany (8):
  - Universitätsklinikum Benjamin Franklin, Berlin, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Lungenklinik Hemer, Hemer
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
  - Pius-Hospital, Oldenburg, Oldenburg
  - National Taiwan University Hospital, Taipei
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Hungary (3):
  - Szent György Hospital, Szekesfehervar, Székesfehérvár
  - Markusovszky County Hospital, Szombathely, Szombathely
  - Zala County Hospital, Zalaegerszeg, Zalaegerszeg
- St James's Hospital, Dublin, Ireland
- Italy (4):
  - Ospedale San Donato di Arezzo, Arezzo
  - Az. USL 4 di Prato, Prato
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Osp. Silvestrin, Sant'Andrea Delle Fratte (PG)
- Japan (16):
  - National Hospital Organization Nagoya Medical Center, Aichi, Nagoya
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - National Hospital Organization Shikoku Cancer Center, Ehime, Matsuyama
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Institute of Biomedical Research and Innovation Hospital, Hyogo, Kobe
  - Kanazawa University Hospital, Ishikawa, Kanazawa
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kurashiki Central Hospital, Okayama, Kurashiki
  - Okayama University Hospital, Okayama, Okayama
  - Kindai University Hospital, Osaka, Osaka-Sayama
  - Osaka City Hospital Organization Osaka City General Hospital, Osaka, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai, Osaka
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
- Malaysia (3):
  - Hospital Pulau Pinang, Palau Pinang
  - Pusat Perubatan University Kebangsaan Malaysia, Wilayah Persekutuan
  - University Malaya Medical Centre, Wilayah Persekutuan
- Peru (3):
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria
  - Clínica Anglo Americana, San Isidro
  - Instituto Nacional de Enfermedades Neoplásicas, Surquillo
- Philippines (3):
  - Perpetual Succour Hospital (Cebu), Cebu City
  - Makati Medical Center, Makati City
  - St. Luke Medical Centre, Quezon
- Romania (2):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - ONCOLAB SRL, Craiova, Craiova
- Russia (6):
  - Republic Clinical Oncology Dispensary, Dept. Chemotherapy, Kazan'
  - FSBSI "N.N Blokhin Medical Research Center of Oncology", Moscow
  - Medical Radiology Science Centre, Obninsk
  - First Pavlov State Medical University Saint Petersburg, Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - FSBI "N.N. Petrov National Medical Research Center of Oncology" of MoH of RF, Saint Petersburg
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - Taipe Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital(TaoYuan), Taoyuan District
- Thailand (4):
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khonkaen
  - Songklanagarind Hospital, Songkhla
- Ukraine (4):
  - City Clinical Hospital #4, Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Donetsk Regional Antitumor Centre, Donetsk
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Lviv State Oncological Regional Treatment & Diagnostic CTR, Lviv
- United Kingdom (7):
  - Royal Devon and Exeter Hospital, Exeter
  - Royal Surrey County Hospital, Guildford
  - The Royal Marsden Hospital, London
  - Maidstone Hospital, Kent Oncology Centre, Maidstone
  - Scunthorpe General Hospital, Oncology, Scunthorpe
  - The Royal Marsden Hospital, Sutton
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III Study of Afatinib or Cisplatin Plus Pemetrexed in Patients With Metastatic Lung Adenocarcinoma With EGFR Mutations. J Clin Oncol. 2023 Jun 1;41(16):2869-2876. doi: 10.1200/JCO.22.02547. PMID 37235976
- [Derived] Wu YL, Sequist LV, Tan EH, Geater SL, Orlov S, Zhang L, Lee KH, Tsai CM, Kato T, Barrios CH, Schuler M, Hirsh V, Yamamoto N, O'Byrne K, Boyer M, Mok T, Peil B, Marten A, Chih-Hsin Yang J, Paz-Ares L, Park K. Afatinib as First-line Treatment of Older Patients With EGFR Mutation-Positive Non-Small-Cell Lung Cancer: Subgroup Analyses of the LUX-Lung 3, LUX-Lung 6, and LUX-Lung 7 Trials. Clin Lung Cancer. 2018 Jul;19(4):e465-e479. doi: 10.1016/j.cllc.2018.03.009. Epub 2018 Mar 17. PMID 29653820
- [Derived] Yang JC, Sequist LV, Zhou C, Schuler M, Geater SL, Mok T, Hu CP, Yamamoto N, Feng J, O'Byrne K, Lu S, Hirsh V, Huang Y, Sebastian M, Okamoto I, Dickgreber N, Shah R, Marten A, Massey D, Wind S, Wu YL. Effect of dose adjustment on the safety and efficacy of afatinib for EGFR mutation-positive lung adenocarcinoma: post hoc analyses of the randomized LUX-Lung 3 and 6 trials. Ann Oncol. 2016 Nov;27(11):2103-2110. doi: 10.1093/annonc/mdw322. Epub 2016 Sep 6. PMID 27601237
- [Derived] Schuler M, Wu YL, Hirsh V, O'Byrne K, Yamamoto N, Mok T, Popat S, Sequist LV, Massey D, Zazulina V, Yang JC. First-Line Afatinib versus Chemotherapy in Patients with Non-Small Cell Lung Cancer and Common Epidermal Growth Factor Receptor Gene Mutations and Brain Metastases. J Thorac Oncol. 2016 Mar;11(3):380-90. doi: 10.1016/j.jtho.2015.11.014. Epub 2016 Jan 25. PMID 26823294
- [Derived] Kato T, Yoshioka H, Okamoto I, Yokoyama A, Hida T, Seto T, Kiura K, Massey D, Seki Y, Yamamoto N. Afatinib versus cisplatin plus pemetrexed in Japanese patients with advanced non-small cell lung cancer harboring activating EGFR mutations: Subgroup analysis of LUX-Lung 3. Cancer Sci. 2015 Sep;106(9):1202-11. doi: 10.1111/cas.12723. Epub 2015 Jul 25. PMID 26094656
- [Derived] Yang JC, Sequist LV, Geater SL, Tsai CM, Mok TS, Schuler M, Yamamoto N, Yu CJ, Ou SH, Zhou C, Massey D, Zazulina V, Wu YL. Clinical activity of afatinib in patients with advanced non-small-cell lung cancer harbouring uncommon EGFR mutations: a combined post-hoc analysis of LUX-Lung 2, LUX-Lung 3, and LUX-Lung 6. Lancet Oncol. 2015 Jul;16(7):830-8. doi: 10.1016/S1470-2045(15)00026-1. Epub 2015 Jun 4. PMID 26051236
- [Derived] Yang JC, Wu YL, Schuler M, Sebastian M, Popat S, Yamamoto N, Zhou C, Hu CP, O'Byrne K, Feng J, Lu S, Huang Y, Geater SL, Lee KY, Tsai CM, Gorbunova V, Hirsh V, Bennouna J, Orlov S, Mok T, Boyer M, Su WC, Lee KH, Kato T, Massey D, Shahidi M, Zazulina V, Sequist LV. Afatinib versus cisplatin-based chemotherapy for EGFR mutation-positive lung adenocarcinoma (LUX-Lung 3 and LUX-Lung 6): analysis of overall survival data from two randomised, phase 3 trials. Lancet Oncol. 2015 Feb;16(2):141-51. doi: 10.1016/S1470-2045(14)71173-8. Epub 2015 Jan 12. PMID 25589191
- [Derived] Yang JC, Hirsh V, Schuler M, Yamamoto N, O'Byrne KJ, Mok TS, Zazulina V, Shahidi M, Lungershausen J, Massey D, Palmer M, Sequist LV. Symptom control and quality of life in LUX-Lung 3: a phase III study of afatinib or cisplatin/pemetrexed in patients with advanced lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3342-50. doi: 10.1200/JCO.2012.46.1764. Epub 2013 Jul 1. PMID 23816967
- [Derived] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-arm, randomised (2:1 ratio), open-label, active-controlled, parallel-group comparison. 345 patients were randomised, 5 patients were not treated: 4 patients were not eligible for treatment and 1 patient in the chemotherapy arm refused to take study medication.
Groups:
- Afatinib 40 mg: Patients received Afatinib monotherapy 40 mg film-coated tablets orally once daily.
- Pemetrexed/Cisplatin Chemotherapy: Patients received Pemetrexed 500 mg/m^2 lyophilised powder as intravenous infusion after Cisplatin 75 mg/m^2 solution for infusion as intravenous infusion on Day 1 of each 21-day treatment course up to 6 cycles.
Period: Overall Study
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Started | 230 (Treated patients.) | 115 (Treated patients.)
Completed | 0 (On treatment at the cut-off date 17MAR2017.) | 0
Not Completed | 230 | 115
Not completed — Progressive disease | 188 | 19
Not completed — Completed 6 courses of chemotherapy | 0 | 60
Not completed — Other Adverse Event (AE) | 28 | 17
Not completed — Protocol Violation | 1 | 4
Not completed — Refusal to continue medication | 7 | 11
Not completed — Not treated | 1 | 4
Not completed — Other not specified above | 5 | 0

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): The randomised set includes all patients who were randomised to receive treatment, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy | Total
Number analyzed (Participants) | 230 | 115 | 345
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (10.1) | 59.9 (10.0) | 60.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 77 | 224
  Male | 83 | 38 | 121
Race/Ethnicity, Customized [Number; unit: Participants] — Race (Asian/non-Asian) was a stratification factor.
  Participants
    Asian | 166 | 83 | 249
    Non-Asian | 64 | 32 | 96
Epidermal Growth Factor Receptor (EGFR) mutation group [Number; unit: Participants] — EGFR mutation group (L858R/Deletion Exon 19/Other) was a stratification factor.
  Participants
    EGFR mutation category: L858R | 91 | 47 | 138
    EGFR mutation category: Deletion Exon 19 | 112 | 57 | 169
    EGFR mutation category: Other | 27 | 11 | 38
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: Participants] — ECOG PS measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction.
  1. Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work.
  2. Ambulatory (>50 percent of waking hours), capable of all self-care, unable to carry out any work activities.
  3. Capable of only limited self-care, confined to bed or chair more than 50 percent of waking hours.
  4. Completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  5. Dead.
  Participants
    ECOG PS 0 (baseline) | 92 | 41 | 133
    ECOG PS 1 (baseline) | 138 | 73 | 211
    ECOG PS 2 (baseline) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Time
Description: PFS was defined as time from randomisation to disease progression or death whichever occured first. Assessed by central independent review according to the Response Evaluation Criteria in Solid Tumours (RECIST 1.1). Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Tumour assessments were performed at Screening, Week 6, Week 12, Week 18 and then every 12-18 weeks until disease progression
Population: Randomised set (RS)
Measure: Median (95% Confidence Interval); unit: Months.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Months. | 11.17 [9.63 to 13.70] | 6.90 [5.39 to 8.25]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0002, Log Rank — Two-sided p-value from log-rank test stratified by EGFR mutation group and race
Statistical Analysis 2: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0002, Regression, Cox; Cox Proportional Hazard (PH) regression stratified by epidermal growth factor receptor (EGFR) mutation group and race; Hazard Ratio (HR) = 0.576, 95% CI [0.426 to 0.778] — Afatinib 40 mg versus Pemetrexed/Cisplatin Chemotherapy

2. Secondary Outcome: Percentage of Patients With Objective Response (OR)
Description: OR was defined as Complete Response (CR) or Partial Response (PR). Assessed by central independent review according to RECIST 1.1.
Time Frame: as for outcome 1
Population: RS.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with OR.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Percentage of patients with OR. | 56.5 [49.8 to 63.0] | 22.6 [15.3 to 31.3]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression stratified for EGFR mutation group and race; Odds Ratio (OR) = 4.802, 95% CI [2.855 to 8.075] — Afatinib 40 mg-Pemetrexed/Cisplatin Chemotherapy

3. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: DC was defined as a patient with OR or Stable Disease (SD). Assessed by central independent review according to the RECIST 1.1.
Time Frame: as for outcome 1
Population: RS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with DC.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Percentage of participants with DC. | 90.4 [85.9 to 93.9] | 80.9 [72.5 to 87.6]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0118, Regression, Logistic; Logistic regression stratified for EGFR mutation group and race; Odds Ratio (OR) = 2.288, 95% CI [1.202 to 4.356] — Afatinib 40 mg-Pemetrexed/Cisplatin Chemotherapy

4. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as time from randomisation to death.
Time Frame: From randomisation to cut-off date (17MAR2017).
Population: RS.
Measure: Median (95% Confidence Interval); unit: Months.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Months. | 28.16 [24.64 to 33.58] | 28.22 [20.73 to 33.22]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.7916, Log Rank — Two-sided p-value from log-rank test stratified by EGFR mutation group and race
Statistical Analysis 2: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.3850, Regression, Cox; Cox PH regression stratified by EGFR mutation group and race; Hazard Ratio (HR) = 0.880, 95% CI [0.660 to 1.174] — Afatinib 40 mg-Pemetrexed/Cisplatin Chemotherapy

5. Secondary Outcome: Tumour Shrinkage
Description: Tumour shrinkage was calculated as the minimum Sum of Diameters (SoD) of target lesions from all post-baseline tumour assessments, as read by the central independent review. The mean of these minimum values were presented after adjusting for baseline SoD, EGFR mutation group and race.
Time Frame: as for outcome 1
Population: RS. There were only 203 patients in the Afatinib 40 mg arm and 101 patients in the Pemetrexed/Cisplatin Chemotherapy with tumour measurements.
Measure: Mean (Standard Error); unit: mm.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 203 | 101
mm. | 33.19 (1.12) | 43.00 (1.59)
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for baseline SoD, EGFR mutation group and race; Mean Difference (Final Values) = -9.82, 95% CI [-13.64 to -5.99] — Afatinib 40 mg-Pemetrexed/Cisplatin Chemotherapy

6. Secondary Outcome: Change From Baseline in Body Weight
Description: Because the PFS was longer for patients in the Afatinib arm than for patients in the chemotherapy arm, the period of data collection for ECOG status and body weight continued for a longer time in the Afatinib arm.
Time Frame: Baseline and throughout the trial until progression (every 3 weeks), up to 28 months.
Population: RS. Only patients with baseline and at least one post-baseline assessment were included.
Measure: Mean (Standard Deviation); unit: Kg.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 224 | 109
Kg.
  Change from baseline at lowest value | -3.95 (3.91) | -2.68 (2.90)
  Change from baseline at last value | -1.19 (5.36) | -0.29 (4.02)

7. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction.
  1. Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work.
  2. Ambulatory (>50 percent of waking hours), capable of all self-care, unable to carry out any work activities.
  3. Capable of only limited self-care, confined to bed or chair more than 50 percent of waking hours.
  4. Completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  5. Dead.
Time Frame: Throughout the trial until progression (every 3 weeks), up to 28 months.
Population: RS. Only patients with baseline and at least one post-baseline assessment were included.
Measure: Number; unit: Participants
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 228 | 111
Participants
  ECOG PS 0 (last value) | 92 | 41
  ECOG PS 1 (last value) | 138 | 73
  ECOG PS 2 (last value) | 0 | 1

8. Secondary Outcome: Health Related Quality of Life (HRQOL): Time to Deterioration in Coughing
Description: HRQOL was measured by European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire C30 (QLQ-C30) and its lung cancer specific module LC13 (QLQ-LC13). Analysis for cough is based on QLQ-LC13 question 1. Time to deterioration was defined as the time from randomisation to a score increased (worsened) by at least 10 points from baseline (0-100 point scale). Patients were considered deteriorated at time of death. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Throughout the trial until progression (every 3 weeks).
Population: RS.
Measure: Median (95% Confidence Interval); unit: Months.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Months. | 26.97 [19.22 to NA] — As only 82 patients (35.7 percent) in the Afatinib 40 mg deteriorated, the upper limit of Confidence Interval (CI) was not estimable. | 8.02 [4.44 to NA] — As only 44 patients (38.3 percent) in the Pemetrexed/Cisplatin Chemotherapy deteriorated, the upper limit of the CI was not estimable.
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0062, Log Rank — Two-sided p-value from log-rank test stratified by EGFR mutation group and race
Statistical Analysis 2: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.2133, Regression, Cox; Cox PH regression stratified by EGFR mutation group and race; Hazard Ratio (HR) = 0.589, 95% CI [0.401 to 0.866] — Afatinib 40 mg vs. Pemetrexed/Cisplatin Chemotherapy, if HR<1 then favours Afatinib 40 mg

9. Secondary Outcome: HRQOL: Time to Deterioration in Dyspnoea
Description: HRQOL was measured by EORTC QLQ-C30 and its lung cancer specific module QLQ-LC13. Analysis for dyspnoea is based on composite of QLQ-LC13 questions 3-5. Time to deterioration was defined as the time from randomisation to a score increased (worsened) by at least 10 points from baseline (0-100 point scale). Patients were considered deteriorated at time of death. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Throughout the trial until progression (every 3 weeks).
Population: RS.
Measure: Median (95% Confidence Interval); unit: Months.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Months. | 10.41 [5.59 to 15.93] | 2.86 [2.17 to 4.90]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0129, Log Rank — Two-sided p-value from log-rank test stratified by EGFR mutation group and race
Statistical Analysis 2: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0078, Regression, Cox; Cox PH regression stratified by EGFR mutation group and race; Hazard Ratio (HR) = 0.680, 95% CI [0.499 to 0.927] — Afatinib 40 mg vs. Pemetrexed/Cisplatin Chemotherapy, if HR<1 then favours Afatinib 40 mg

10. Secondary Outcome: HRQOL: Time to Deterioration in Pain
Description: HRQOL was measured by EORTC QLQ-C30 and its lung cancer specific module QLQ-LC13. Analysis for pain is based on composite of QLQ-C30 questions 9 and 19. Time to deterioration was defined as the time from randomisation to a score increased (worsened) by at least 10 points from baseline (0-100 point scale). Patients were considered deteriorated at time of death. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Throughout the trial until progression (every 3 weeks).
Population: RS.
Measure: Median (95% Confidence Interval); unit: Months.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Number analyzed (Participants) | 230 | 115
Months. | 4.17 [2.79 to 5.59] | 3.09 [2.17 to 3.98]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.1882, Log Rank — Two-sided p-value from log-rank test stratified by EGFR mutation group and race
Statistical Analysis 2: Comparison: Afatinib 40 mg vs Pemetrexed/Cisplatin Chemotherapy; Test type: Superiority or Other; p = 0.0427, Regression, Cox; Cox PH regression stratified by EGFR mutation group and race; Hazard Ratio (HR) = 0.826, 95% CI [0.618 to 1.104] — Afatinib 40 mg vs. Pemetrexed/Cisplatin Chemotherapy, if HR<1 then favours Afatinib 40 mg

11. Secondary Outcome: Trough Plasma Concentrations of Afatinib at Day 22
Description: Trough plasma concentrations of Afatinib at Day 22 (course 2, visit 1) after multiple daily dosing of 40 mg Afatinib and after dose escalation to 50 mg or dose reduction to 30 mg or 20 mg.
Time Frame: Day 22.
Population: Patients from the treated set with evaluable data and who had at least 1 valid Afatinib plasma concentration available on this time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL.
Groups:
- Afatinib 20 mg: Patients received Afatinib monotherapy 20 mg film-coated tablets orally once daily after a dose reduction.
- Afatinib 30 mg: Patients received Afatinib monotherapy 30 mg film-coated tablets orally once daily after a dose reduction.
- Afatinib 50 mg: Patients received Afatinib monotherapy 50 mg film-coated tablets orally once daily after a dose escalation.
Arm/Group | Afatinib 20 mg | Afatinib 30 mg | Afatinib 40 mg | Afatinib 50 mg
Number analyzed (Participants) | 0 | 11 | 165 | 3
ng/mL. |  | 21.8 (36.6) | 28.0 (85.0) | 29.9 (46.1)

12. Secondary Outcome: Trough Plasma Concentrations of Afatinib at Day 29
Description: Trough plasma concentrations of Afatinib at day 29 (course 2, visit 2) after multiple daily dosing of 40 mg Afatinib and after dose escalation to 50 mg or dose reduction to 30 mg or 20 mg.
Time Frame: Day 29.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL.
Arm/Group | Afatinib 20 mg | Afatinib 30 mg | Afatinib 40 mg | Afatinib 50 mg
Number analyzed (Participants) | 0 | 25 | 143 | 16
ng/mL. |  | 28.0 (82.4) | 25.8 (69.5) | 29.6 (79.2)

13. Secondary Outcome: Trough Plasma Concentrations of Afatinib at Day 43
Description: Trough plasma concentrations of Afatinib at Day 43 (course 3, visit 1) after multiple daily dosing of 40 mg Afatinib and after dose escalation to 50 mg or dose reduction to 30 mg or 20 mg.
Time Frame: Day 43.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL.
Arm/Group | Afatinib 20 mg | Afatinib 30 mg | Afatinib 40 mg | Afatinib 50 mg
Number analyzed (Participants) | 2 | 39 | 126 | 14
ng/mL. | 24.4 (260) | 24.7 (63.9) | 23.5 (66.2) | 27.5 (64.4)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication.
Arm/Group | Afatinib 40 mg | Pemetrexed/Cisplatin Chemotherapy
Serious Adverse Events (participants affected / at risk) | 72/229 | 25/111
Other Adverse Events (participants affected / at risk) | 229/229 | 108/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=229) | Pemetrexed/Cisplatin Chemotherapy (N=111)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 11 | 3
Abasia (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Death (General disorders) | 2 | 1
Disease progression (General disorders) | 2 | 0
Fatigue (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 1 | 1
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Schizophreniform disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=229) | Pemetrexed/Cisplatin Chemotherapy (N=111)
Anaemia (Blood and lymphatic system disorders) | 19 | 29
Leukopenia (Blood and lymphatic system disorders) | 6 | 21
Neutropenia (Blood and lymphatic system disorders) | 4 | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 8
Dry eye (Eye disorders) | 14 | 0
Vision blurred (Eye disorders) | 12 | 2
Abdominal pain (Gastrointestinal disorders) | 13 | 5
Abdominal pain upper (Gastrointestinal disorders) | 15 | 8
Cheilitis (Gastrointestinal disorders) | 22 | 0
Constipation (Gastrointestinal disorders) | 37 | 39
Diarrhoea (Gastrointestinal disorders) | 216 | 25
Dyspepsia (Gastrointestinal disorders) | 21 | 7
Mouth ulceration (Gastrointestinal disorders) | 24 | 3
Nausea (Gastrointestinal disorders) | 65 | 75
Stomatitis (Gastrointestinal disorders) | 88 | 10
Vomiting (Gastrointestinal disorders) | 53 | 50
Asthenia (General disorders) | 16 | 14
Chest pain (General disorders) | 16 | 14
Fatigue (General disorders) | 45 | 39
Malaise (General disorders) | 7 | 6
Mucosal inflammation (General disorders) | 67 | 5
Oedema (General disorders) | 7 | 13
Oedema peripheral (General disorders) | 17 | 8
Pyrexia (General disorders) | 28 | 6
Conjunctivitis (Infections and infestations) | 28 | 3
Cystitis (Infections and infestations) | 15 | 1
Folliculitis (Infections and infestations) | 12 | 0
Nasopharyngitis (Infections and infestations) | 39 | 9
Paronychia (Infections and infestations) | 132 | 0
Upper respiratory tract infection (Infections and infestations) | 29 | 4
Urinary tract infection (Infections and infestations) | 19 | 5
Alanine aminotransferase increased (Investigations) | 27 | 3
Aspartate aminotransferase increased (Investigations) | 22 | 1
Blood creatinine increased (Investigations) | 5 | 10
Haemoglobin decreased (Investigations) | 3 | 13
Neutrophil count decreased (Investigations) | 1 | 8
Weight decreased (Investigations) | 44 | 16
Decreased appetite (Metabolism and nutrition disorders) | 70 | 61
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 4
Dizziness (Nervous system disorders) | 28 | 12
Dysgeusia (Nervous system disorders) | 18 | 9
Headache (Nervous system disorders) | 37 | 19
Insomnia (Psychiatric disorders) | 37 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Acne (Skin and subcutaneous tissue disorders) | 52 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 20
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 32 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 72 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 14 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 50 | 1
Rash (Skin and subcutaneous tissue disorders) | 145 | 11
Skin exfoliation (Skin and subcutaneous tissue disorders) | 13 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 16 | 0
Hypertension (Vascular disorders) | 14 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.